CLINICAL TRIAL: NCT06757608
Title: Postprandial Responses to Fish Intake: in Vivo and in Vitro Study
Brief Title: Postprandial Responses to Fish Intake
Acronym: PREFish
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Ministry of Education, Brazil (Other Government)
Responsible Party: Principal Investigator, Jarlei Fiamoncini, Professor PhD, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 69418723.6.0000.0067
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Post-prandial Glycaemic Response; Postprandial Lipids Metabolism; Postprandial Metabolism
Keywords: Cardiovascular diseases; Metabolism; Metabolomics; Fish; Dietary protein
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Crossover Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tambaqui meat (Active Comparator): Tambaqui (Colossoma macropomum) meat intake, 7g per BMI unit
  Interventions: Other: Assessment of postprandial metabolism after intake of different meat
- Sardine meat (Active Comparator): Sardine (Opisthonema oglinum) meat intake, 7g per BMI unit
  Interventions: Other: Assessment of postprandial metabolism after intake of different meat
- Beef (Active Comparator): Beef (Bos taurus) meat intake, 7g per BMI unit
  Interventions: Other: Assessment of postprandial metabolism after intake of different meat

INTERVENTIONS:
Other: Assessment of postprandial metabolism after intake of different meat — 30 healthy adults (15 male and 15 female) consumed sardines (Opisthonema oglinum, marine fish), tambaqui (Colossoma macropomum, freshwater culture), and beef (Bos taurus). The meal consisted only of meat, with 7g per BMI unit. The postprandial response was observed for 5 hours, after an overnight fast.

SUMMARY:
Fish consumption has been increasing in recent decades due to consumer interest in the positive health effects of regular food intake, among other factors. Previous studies have described significant results on the acute consumption of fish products, favoring the reduction of triglycerides, total cholesterol, low-density lipoprotein, reduced insulin secretion, and increased plasma concentration of high-density lipoprotein during the postprandial period. Despite this scenario, studies investigating acute metabolic responses, such as postprandial physiological phenomena after consumption of the main fish species ingested by Brazilians, are still scarce. Thus, investigations of the acute effects of fish intake on postprandial metabolism may reveal new beneficial effects associated with this food group. The present proposal aims to compare the acute effects of the ingestion of two sources of fish and bovine protein on postprandial metabolism through the capillary blood sample collected within 5 hours after the ingestion of test meals, investigating hormones and inflammatory mediators and quantifying triglycerides, total cholesterol and non-esterified fatty acids and blood glucose, in addition to evaluating sensory aspects and satiety between different meals. It is expected to generate new data on postprandial physiology and investigate possible effects of fish ingestion that can contribute to public health management and healthy eating patterns.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 35 years and with a body mass index between 20 and 29 kg/m2.

Exclusion Criteria:

* Individuals with a vegetarian/vegan diet, a history of fish allergy, aversion to fish, used supplementation with n-3 polyunsaturated fatty acids or probiotics, who have a diagnosis of pregnancy, dyslipidemia, diabetes, inflammatory bowel disease, liver disease, who have undergone surgeries that alter the anatomy of the digestive tract (bariatric surgery or cholecystectomy, for example) and use of antimicrobial therapy in the 3 months before the study will not be allowed to participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma markers of intermediate metabolism and inflammation | 3 weeks
  Capillary blood samples (approximately 500 µL) were collected after a 12-hour fasting and in different time points within a 5-hours interval after food intake to assess plasma metabolic and inflammatory markers (cytokines), aiming at identifying their response to the food intake.

SECONDARY OUTCOMES:
Urine metabolome | 3 weeks
  Urine samples were collected after a 12-hours fasting and during the postprandial period (all urine produced during the first 5 hours following food intake) to assess changes in urinary metabolome induced by the intake of the tested meal.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No